CLINICAL TRIAL: NCT00570427
Title: Improving Depression Treatment for Older Minority Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Isabel T. Lagomasino, MD MSHS, Keck School of Medicine, University of Southern California
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG0091; 5P30AG021684 (NIH); 1557 G GD102
Record Dates: First submitted 2007-12-07; First posted 2007-12-11 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: Depression
Keywords: psychotherapy; behavior therapy; counseling; aging; medically underserved population
MeSH Terms: conditions — Depression | interventions — Medication Therapy Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1. (Experimental): All participants
  Interventions: Behavioral: Problem Solving Therapy (PST); Behavioral: Medication Management

INTERVENTIONS:
Behavioral: Problem Solving Therapy (PST) — Counseling
Behavioral: Medication Management — If a participant chooses to receive antidepressant medication while in the study, a depression care specialist works with the participant's usual primary care provider to initiate an appropriate prescription and to follow-up with side effects, adherence, efficacy, etc. on a monthly or biweekly basis.

SUMMARY:
The purpose of this study is to improve access to quality depression care for older, low-income, minority adults in public sector health care. The study will examine current depression care in a public sector geriatric clinic that serves mostly Spanish-speaking Latinos and pilot study assessments and treatments in order to lay the groundwork for a large study of quality improvement for depressed older minorities

DETAILED DESCRIPTION:
Depressive disorders affect 5-10% of older primary care patients, although rates may be higher among Latinos, especially among immigrants and those less acculturated. Late-life depression may be chronic and recurrent and results in significant morbidity and mortality. Despite a growing evidence base for the treatment of geriatric depression, only half of depressed older adults receive mental health care; fewer than 10% receive specialty services. Treatment rates are even lower for low-income, ethnic minorities who may be more ill and disabled, may lack adequate insurance and have different treatment preferences, and who frequently face barriers to accessing care. Recent quality improvement interventions for geriatric depression have targeted primary care, the location where older patients and ethnic minorities are most likely to receive mental health services. A recent multi-site, randomized trial of collaborative care for geriatric depression in primary care offered patients their choice of treatments, including antidepressant medication or 6-8 sessions of a structured psychotherapy. Although the intervention had few cultural accommodations, both processes and outcomes of care improved for depressed older minorities. However, because the study only included Latinos who were English-speaking and mostly high school graduates, these results may not generalize to a large proportion of ethnic minorities.

This study first examines current rates of depression and patterns of depression treatment in a public-sector geriatric clinic that serves mostly Spanish-speaking Latinos. Then depressed patients are identified and their depression treatment preferences and barriers to care are assessed. Patients are enrolled in a 6-month patient-centered, evidence-based intervention, and they, family members, and clinic medical providers are interviewed at program end to assess the feasibility, acceptability, and possible effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the LAC+USC Medical Center Geriatric Clinic
* English- or Spanish-speaking
* Positive for depression on the Geriatric Depression Scale
* Current major depressive disorder or dysthymia
* All adult family members, especially caregivers, and all regular clinic providers eligible for interviews

Exclusion Criteria:

* History of bipolar disorder or psychosis
* Significant cognitive impairment (score less than 24 on the Mini-Mental Status Examination, adjusted for age and education)
* Acute suicidal ideation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Depression severity, depression treatment preferences, and barriers to care | baseline and 6 months

SECONDARY OUTCOMES:
Feasibility, acceptability, and effectiveness of intervention | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Isabel T. Lagomasino, MD MSHS, Principal Investigator — Department of Psychiatry, Keck School of Medicine, University of Southern California
Locations (1):
- LAC+USC Medical Center Geriatric Clinic, Los Angeles, California, United States

REFERENCES:
- [Background] Dwight-Johnson M, Lagomasino IT. Addressing depression treatment preferences of ethnic minority patients. Gen Hosp Psychiatry. 2007 May-Jun;29(3):179-81. doi: 10.1016/j.genhosppsych.2007.02.001. No abstract available. PMID 17484933
- [Background] Vega WA, Karno M, Alegria M, Alvidrez J, Bernal G, Escamilla M, Escobar J, Guarnaccia P, Jenkins J, Kopelowicz A, Lagomasino IT, Lewis-Fernandez R, Marin H, Lopez S, Loue S. Research issues for improving treatment of U.S. Hispanics with persistent mental disorders. Psychiatr Serv. 2007 Mar;58(3):385-94. doi: 10.1176/ps.2007.58.3.385. PMID 17325113
- [Background] Lagomasino IT, Dwight-Johnson M, Miranda J, Zhang L, Liao D, Duan N, Wells KB. Disparities in depression treatment for Latinos and site of care. Psychiatr Serv. 2005 Dec;56(12):1517-23. doi: 10.1176/appi.ps.56.12.1517. PMID 16339612